CLINICAL TRIAL: NCT01470482
Title: Does Tourniquet Use in Total Knee Replacement Improve Fixation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Per Aspenberg (Other)
Responsible Party: Sponsor-Investigator, Per Aspenberg, Professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ledin01; VR - 2009-6725). (Other: EPN Linköping M59-06)
Record Dates: First submitted 2011-11-03; First posted 2011-11-11 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee; Tourniquet; Blood loss; pain; range of motion
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage; Pain | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Tourniquet (Other): We compare tourniquet or not in knee surgery
  Interventions: Procedure: No use of tourniquet
- Tourniquet (Active Comparator): We compare tourniquet or not in knee surgery
  Interventions: Procedure: Tourniquet

INTERVENTIONS:
Procedure: No use of tourniquet — Tourniquet is not applied i 25 pts
  Other Names: No Tourniquet
  Arms: No Tourniquet
Procedure: Tourniquet — Use of tourniquet
  Arms: Tourniquet

SUMMARY:
Although a tourniquet may reduce bleeding during total knee replacement (TKA), and thereby improve fixation, it might also cause complications. Migration as measured by RadioStereometric Analysis (RSA) can predict future loosening. We will investigate if the use of a tourniquet influences fixation measured with RSA.

DETAILED DESCRIPTION:
The use of a tourniquet during total knee replacement (TKA) is a generally accepted routine at many departments. It is thought to facilitate dissection and reduce peroperative bleeding, but the main argument for its use is that bleeding bone surfaces might impair the fixation of cemented prostheses, because of less cement penetration.

We investigate in a RCT 50 patient with radiostereometric analysis, where 25 is randomized to a tourniquet during the hole operation and 25 are not.

Primary outcome is MTPM, a meassure of migration(loosening) of the kneeprosthesis.

Secondary outcomes are total bleeeding, pain, range of motion and outcome of a patient self assesed knee score (KOOS) Total follow up time 2 years

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary osteoarthritis without other severe disease (ASA 1-2).

Exclusion Criteria:

* were inability to give informed consent,
* rheumatic arthritis,
* malignancy,
* coagulation disorder or medical treatment influencing the coagulation,
* liver disease,
* severe heart disease or bilateral operation.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
View protocol record | 2 years
  Measures the migration of the knee prosthesis

SECONDARY OUTCOMES:
View Protocol Record | 2 years
  Meassures of total bledding, ROM, KOOS, Pain

CONTACTS AND LOCATIONS:
Overall Officials: Per Aspenberg, MD,PhD, Study Director — Linkoeping University
Locations (1):
- Motala hospital, Motala, Sweden